CLINICAL TRIAL: NCT03794115
Title: Differential Expression of Immune Repertoire of T/B Lymphocytes in Ovarian High Grade Serous Carcinoma
Brief Title: Immune Repertoire of Ovarian HGSC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: EOC-IMMUNE
Record Dates: First submitted 2019-01-03; First posted 2019-01-04 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Ovarian High Grade Serous Carcinoma; Immune Repertoire; T Lymphocyte Receptor; B Lymphocyte Receptor
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood and carcinoma tissue with pericarcinomatous tissue are taken from the patients with ovarian high grade serous carcinoma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Treatment for ovarian cancer — The treatment for ovarian cancer includes the debulking surgery and platinum-based chemotherapy.

SUMMARY:
In this preliminary study, peripheral blood and carcinoma tissue with pericarcinomatous tissue are taken from the patients with ovarian high grade serous carcinoma at several points: before any treatment, after the debulking surgery, and after all the proposed chemotherapy. The differential expression of the T/B lymphocyte receptors in these samples will be analyzed with the platinum-based treatment and survival outcomes of the patients. The primary objective is the expression rates of T/B lymphocyte receptors in different stages of checking points.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed of primary ovarian high grade serous carcinoma
* Aged 18 years or older
* No immunosuppressive disease
* Signed an approved informed consents

Exclusion Criteria:

* Not meeting all of the inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients confirmed of primary ovarian high grade serous carcinoma, aged 18 years or older and accept systematic treatment including debulking surgery and platinum-based chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-01-03 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Expression rates of T lymphocyte receptors | One year
  Expression rates of T lymphocyte receptors in different stages of checking points, including timings before any treatment, after the debulking surgery, and after all the proposed chemotherapy
Expression rates of B lymphocyte receptors | One year
  Expression rates of T lymphocyte receptors in different stages of checking points, including timings before any treatment, after the debulking surgery, and after all the proposed chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided